CLINICAL TRIAL: NCT06964256
Title: Evaluation of the Efficacy and Safety of sEMG Monitoring of Lower Abdominal Breathing Training in the Treatment of Urinary Retention After Spinal Cord Injury: a Randomized Controlled Trial
Brief Title: Clinical Trial of Abdominal Breathing for Urinary Retention After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYLL_202404_001
Record Dates: First submitted 2025-04-17; First posted 2025-05-09 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries (SCI); Urinary Retention
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Retention | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: conventional rehabilitation treatment. (Active Comparator): Conventional rehabilitation treatment methods include intermittent catheterization and acupuncture. Intermittent catheterization is based on the results of urodynamic examination to develop a personalized drinking plan and the number of catheterization, and the number of catheterization is selected according to the amount of residual urine; Intermittent catheterization can reduce the rate of urinary tract infections, the incidence of urethral stones, and improve bladder capacity. Acupuncture treatment improves the patient's urinary function by acupuncture on the lower abdomen and lumbosacral acupoints once a day, 5 days a week, for a total of 3 weeks
  Interventions: Other: Control group: intermittent catheterization; Other: Control group and experimental group: acupuncture treatment
- Experimental group: Conventional rehabilitation treatment sEMG monitoring of lower abdominal breathi (Experimental): Experimental group: Conventional rehabilitation treatment sEMG monitoring of lower abdominal breathing training.
  The conventional rehabilitation treatment method is the same as above; The specific operation of sEMG abdominal breathing training: ask the patient to empty the bladder before training, the patient to take a supine position, hip and knee flexion 60 degrees (for those who cannot maintain hip and knee flexion in the lower limbs, family members can assist), at the same time, the electrodes are attached to both sides of the patient's anus, the reference electrode is attached to the anterior superior iliac spine, the biostimulation feedback instrument is used to collect the patient's pelvic floor muscle electromyography value, and the patient is instructed to breathe in the abdomen, slowly inhale through the nose when inhaling, and put the hand on the abdomen to feel the abdomen slowly bulge for 3-5s; Exhale slowly with your mouth and slowly tighten your abdomen for 3-5s; For p
  Interventions: Behavioral: Abdominal breathing exercises; Behavioral: Experimental group: intermittent catheterization; Other: Control group and experimental group: acupuncture treatment

INTERVENTIONS:
Behavioral: Abdominal breathing exercises — Control group: conventional rehabilitation treatment. Conventional rehabilitation treatment methods include intermittent catheterization and acupuncture. Intermittent catheterization is based on the results of urodynamic examination to develop a personalized drinking plan and the number of catheterization, and the number of catheterization is selected according to the amount of residual urine; Intermittent catheterization can reduce the rate of urinary tract infections, the incidence of urethral stones, and improve bladder capacity. Acupuncture treatment improves the patient's urinary function by acupuncture on the lower abdomen and lumbosacral acupoints once a day, 5 days a week, for a total of 3 weeks Experimental group: Conventional rehabilitation treatment sEMG monitoring of lower abdominal breathing training.
  The conventional rehabilitation treatment method is the same as above; The specific operation of sEMG abdominal breathing training: ask the patient to empty the bladder befor
  Arms: Experimental group: Conventional rehabilitation treatment sEMG monitoring of lower abdominal breathi
Other: Control group: intermittent catheterization — Intermittent catheterization is based on the results of urodynamic examination to develop a personalized drinking plan and the number of catheterization, and the number of catheterization is selected according to the amount of residual urine; Intermittent catheterization can reduce the rate of urinary tract infections, the incidence of urethral stones, and improve bladder capacity. Acupuncture treatment improves the patient's urinary function by acupuncture on the lower abdomen and lumbosacral acupoints once a day, 5 days a week, for a total of 3 weeks
  Other Names: Control group: Acupuncture treatment
  Arms: Control group: conventional rehabilitation treatment.
Behavioral: Experimental group: intermittent catheterization — Conventional rehabilitation treatment methods include intermittent catheterization and acupuncture. Intermittent catheterization is based on the results of urodynamic examination to develop a personalized drinking plan and the number of catheterization, and the number of catheterization is selected according to the amount of residual urine; Intermittent catheterization can reduce the rate of urinary tract infections, the incidence of urethral stones, and improve bladder capacity. Acupuncture treatment improves the patient's urinary function by acupuncture on the lower abdomen and lumbosacral acupoints once a day, 5 days a week, for a total of 3 weeks. The specific operation of sEMG abdominal breathing training: ask the patient to empty the bladder before training, the patient to take a supine position, hip and knee flexion 60 degrees (for those who cannot maintain hip and knee flexion in the lower limbs, family members can assist), at the same time, the electrodes are attached to both
  Other Names: Experimental group: acupuncture treatment; Experimental group: abdominal breathing training
  Arms: Experimental group: Conventional rehabilitation treatment sEMG monitoring of lower abdominal breathi
Other: Control group and experimental group: acupuncture treatment — Acupuncture treatment uses acupuncture to act on the acupuncture points in the lower abdomen and lumbosacral region to improve the patient's urination function

SUMMARY:
Randomized controlled trials were conducted in patients with urinary retention after spinal cord injury. The effects of abdominal breathing training on pelvic floor muscle tone, muscle strength and residual urine volume in patients with urinary retention after spinal cord injury were observed by Glazer and bladder volume measurement to compare the electromyography value and residual urine volume of pelvic floor muscles at different stages of resting state and contraction state of the two groups, and the subjective feelings of the patients were evaluated in combination with relevant scales. To provide a scientific basis for abdominal breathing as an adjuvant treatment for urinary retention after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:(1) Meet the "International Standards for the Neurological Classification of Spinal Cord Injuries" formulated by the American Spinal Cord Injury Association, and after the end of the spinal cord shock period, the ASIA classification is B, C, and D, and the clinical manifestations are urinary retention, residual urine > 100ml, and gender is not limited; (2) Age 16-80 years old; (3) The course of the disease is within 12 months; (4) Intermittent catheterization; (5) Pelvic floor muscle function test shows pelvic floor muscle hypotonia; (6) Have good communication skills, voluntarily participate in the trial and sign the informed consent form.

-

Exclusion Criteria:

(1) Patients with severe urinary tract infection and hydronephrosis; (2) Those with other serious diseases; (3) Respiratory failure or tracheostomy; (4) patients with urinary retention not caused by spinal cord injury; (5) Dermato-electrode passers; (6) Patients with consciousness impairment and cognitive impairment; (7) Patients with poor treatment compliance and inability to follow doctor's instructions.

-

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Bladder residual urine output at 3 weeks | Three weeks
  A bladder volume measuring instrument (model HD5, produced by Liaoning Hande Technology Co., Ltd.) was used to perform ultrasound detection and record the residual urine volume after urination.

SECONDARY OUTCOMES:
Glazer assessment value | Three weeks
  Pelvic floor biostimulation feedback instrument Glazer evaluation was used to compare the resting state and contraction state of the two groups of patients at different stages of pelvic floor muscle electromyography
Short-form Health Survey-Qualiveen | Three weeks
  The scale includes 4 dimensions and 8 items of annoyance (items 1~2), restriction (items 3~4), fear (items 5~6), and feeling (items 7~8). Each item was scored by Likert 5 grades, in which item 3 was assigned a score of "never", "rarely", "sometimes", "often" and "always", and the rest of the items were assigned 0~4 points according to "none", "a little", "moderate", "quite severe" and "extremely severe", the score of each dimension was the mean of each item within the dimension, and the score of the scale was the average score of each dimension, with a total score of 0~4 points, the lower the score, the better the quality of life of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- 107 Wenhua Xi Road, Ji'nan Shandong 250012, Jinan, jinan, China

IPD SHARING:
Plan to Share IPD: No